CLINICAL TRIAL: NCT02477202
Title: Mirena® IUD's Effect on Fallopian Tube Fimbriae and Ovarian Cortical Inclusion Cyst Cell Proliferation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-105
Record Dates: First submitted 2015-06-15; First posted 2015-06-22 (Estimated); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-01

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Mirena® IUD's; Women; risk-reducing salpingo-oophorectomy; risk-reducing salpingectomy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

ARMS (1):
- Mirena® IUD (Experimental): This is a non-randomized study of the effect of Mirena® IUD use of at least 10 days before an RRSO or RRS on cell proliferation within the FTF and when available within ovarian CICs in women aged 35 through 50. The study will compare the results from 14 women using Mirena® with the results from 28 normally cycling women identified under MSK IRB Protocol #14-165 described above; all patients will be aged 35-50 years, and will have undergone the RRSO at MSK. To date we have identified approximately 100 suitable controls and are continuing to identify further suitable controls among women who have recently undergone RRSOs at MSK. The balancing/matching factors will be BRCA status (BRCA1/BRCA2/BRCA-ve), age (35-39/40-44/45-50), parity (nulliparous/parous), and BMI (<30/30+ kg/m^2). As each Mirena® patient completes the study and is deemed evaluable, she will be matched on each of these factors with 2 controls.
  Interventions: Device: Mirena® intra-uterine device (IUD)

INTERVENTIONS:
Device: Mirena® intra-uterine device (IUD) — In this study, a Mirena® IUD will be inserted into volunteers scheduled for a risk-reducing salpingo-oophorectomy (RRSO) or risk-reducing salpingectomy (RRS) at Memorial Sloan Kettering Cancer Center (MSK). Alternatively, women with a Mirena® IUD already in place and who will be scheduled for an RRSO or RRS at MSK can also participate. We are seeking 14 evaluable participants. FTF tissue (and ovarian inclusion cyst tissue, when available) collected at the time of risk-reducing salpingectomy (RRS) will be tested by immunochemistry staining for Ki67 (a protein that is significantly increased when cells are preparing for division).

SUMMARY:
Combination-type oral contraceptives (COCs) have been shown to significantly reduce the risk of invasive epithelial ovarian cancer (IEOC); this protective effect may be achieved to a large extent through COCs ability to reduce cell proliferation in the fallopian tube fimbriae (FTF). The progestin-releasing Mirena® intra-uterine device (IUD) is an increasingly popular method of contraception, but it is not known if its use will reduce a woman's risk of IEOC. Mirena® use does not block ovulation in most women but it may release sufficient progestin to also reduce cell proliferation in the FTF. This study aims to evaluate the effects of the Mirena® IUD on cell proliferation in the FTF as a possible biomarker of protection against IEOC.

ELIGIBILITY:
Inclusion Criteria:

* Women between 35 and 50 years of age (inclusive)
* Women who will be scheduled to undergo an RRSO or RRs
* Women who will have at least one fallopian tube removed for risk-reducing reasons (with or without removal of ovar(ies))
* Women who are willing to have a Mirena® IUD inserted at least prior to risk-reducing surgery or who already have the Mirena® in place
* Women using non-hormonal forms of contraception (Note: If a copper IUD is being used, the IUD must be removed prior to or at time of Mirena insertion.)

Exclusion Criteria:

* Any medical contraindication to use of a Mirena® IUD, including:

  * Pregnancy (a pregnancy test is required prior to study entry)
  * Known uterine anomaly that distorts the shape of the uterine cavity
  * Acute pelvic inflammatory disease
  * Postpartum endometritis or endometrial infection
  * Known or suspected uterine or cervical neoplasia
  * Known history or suspected breast cancer or other progestin-sensitive cancer
  * Uterine bleeding of unknown etiology.
  * Untreated acute cervicitis, vaginitis, or other lower genital tract infections
  * Acute liver disease or liver tumor (benign or malignant)
* Use of tamoxifen, raloxifene, or chemotherapy within the previous 6 months
* Positive pregnancy test
* Breastfeeding
* Use of a copper IUD if the patient is not willing to have it removed prior to surgery and replaced with a Mirena® IUD

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirena® IUD: This is a non-randomized study of the effect of Mirena® IUD use of at least 10 days before an RRSO or RRS on cell proliferation within the FTF and when available within ovarian CICs in women aged 35 through 50. The study will compare the results from 14 women using Mirena® with the results from 28 normally cycling women identified under MSK IRB Protocol #14-165 described above; all patients will be aged 35-50 years, and will have undergone the RRSO at MSK. To date we have identified approximately 100 suitable controls and are continuing to identify further suitable controls among women who have recently undergone RRSOs at MSK.
Period: Overall Study
Arm/Group | Mirena® IUD
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mirena® IUD
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 38 [37 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Cell Proliferation in the Fallopian Tube Fimbriae as Measured by Ki-67%+
Description: Women will be deemed evaluable for this primary outcome if they successfully underwent placement of the Mirena® IUD, received a RRSO or RRS as planned, and had a P4 value ≤1 ng/ml.
Time Frame: 1 year
Measure: Median (Full Range); unit: percentage of positively stained cells
Arm/Group | Mirena® IUD
Number analyzed (Participants) | 7
percentage of positively stained cells | 8.3 [0 to 15]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Mirena® IUD
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT02477202/Prot_SAP_000.pdf